CLINICAL TRIAL: NCT03787316
Title: The Effects of Custom-made Insoles on Foot Pressure Redistribution and Spatio - Temporal Gait Parameters in Sever Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATADEK- 2018/13
Record Dates: First submitted 2018-12-13; First posted 2018-12-26 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2019-02

CONDITIONS: Calcaneal Apophysitis; Gait; Sever's Disease
Keywords: gait; sever's

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 4-weeks use of specially produced shock absorbing insoles and the daily home exercise program during this 4 weeks. Daily exercises include M. gastrocnemius, soleus, tibialis anterior, tibialis posterior stretching, strengthening of the anterior, lateral, posterior compartmental and foot intrinsic muscles of the foot, eccentric exercise of gastrocnemius and soleus.
  Interventions: Device: Study group

INTERVENTIONS:
Device: Study group — 4 weeks of custom-made insoles in the home and outside the home environment , follow the home exercise program during this process.It is planned to perform gait parameters and pain assessment before and after the treatment.

SUMMARY:
The aim of this study was to investigate the effect of specially produced insoles on biomechanical and gait parameters in children with Sever's disease.

DETAILED DESCRIPTION:
Introduction: Sever's disease or calcaneal apophysitis is common in pediatric and adolescent patients and characterized by heel pain. Inflammation of apophysis in children of growing age causes microabrasion in bone cartilage joint. At the same time, the disease affects the self-limitation and affects the maturation of calcaneus.Sever's disease is an overuse syndrome and was described by James Warren Sever in 1912. The prevalence of Sever's disease varies between 2% and 16%.Sever's more common in children aged 8 - 15 years, but it was reported that heel pain increased during or after activity.This results in a shortening of the stance phase to remove the limb to avoid heel strikes during walking. Increased tension in the Achilles tendon and plantar fascia is affected by the mobility of the medial longitudinal arch of the foot and increases loading on the calcaneal cartilage. Stimulates foot alignment to pronation.

Different treatment have been described in Sever's disease. In the treatment program, stretching, strengthening exercises and ice application are recommended especially for gastrocnemius muscle and extensor muscle group.The traditional treatment approach is the restriction of the child's physical activity and sporting activities and rest until the symptoms have passed. In addition, orthoses can be used to treat the heel amplifier, anatomical dysregulation dominated by standing pronation. There is no previous study in order to investigate the effect of the specially produced insoles on the Sever's disease by changing the foot pressure center and the effect of the pronation on the gait parameters.

Subjects and methods:

The study is planned to be done with physical examination and radiological imaging of the patients who are between 8 and 15 years of age and diagnosed with Sever's disease. After the first physical examination evaluation, the foot rotation, step length, stance phase percentage, swing phase percentage, cadence and velocity parameters will be recorded with Zebris FDM -T (Force Distribution Measurement Treadmill) system. Zebris is a name of company in Germany.

Zebris Medical Limited ) is an innovative company that has been successful for many years in the development and production of 3D motion analysis and force measurement technologies for biomechanics. When the treadmill is in static and dynamic condition, strong pressure distribution measurement will be taken and personalized insole production according to foot pressure map will be done by orthosis prosthesis technician with Arch drafters Orthotics technology. After physiotherapist,decision, it will be delivered to the patients with the condition of being used outside and inside the home. Measurements related to pressure and gait parameters will be repeated after 4 weeks of use and home exercise (strengthening, stretching and eccentric exercise for the anterior lateral - posterior compartment of the foot ).

The spatio temporal gait parameters of the patients will be evaluated with Zebris (Zebris Medical Limited , Germany) FDM (Force Distribution Measurement ) treadmill system and pain levels at rest and during activity will be questioned using Visual Analog Scale.

Sample size: 40 professional athlete who are between 8 and 15 years of age for experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8-15 years
* Calcaneal apophysitis with clinical symptoms and radiographic screening
* Positive squeeze test sign
* Heel pain more than 2 weeks

Exclusion Criteria:

* Intermittent heel pain to exclude plantar fasciitis pathology
* Another pathology within the same or the other foot for example fracture, achilles tendinitis and calcaneal bursitis
* Another pain symptom within the other part of the extremity

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Step length (centimeter- cm) | 4 weeks
  Step length (cm), will be evaluated by Zebris (Zebris Medical Limited - Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.
Pain - Visual Analogue Scale- | 4 weeks
  Visual Analogue Scale is one of the simple and common methods used in pain assessment. Self reported pain intensity during the rest and the activity measured by 0-10 centimeter chart. Visual Analogue Scale (VAS), where 0 indicates no pain or best and 10 indicates the most intense pain imaginable or worst. The patient will mark the severity of the pain on a 10 cm long chart.
Stride length (centimeter -cm) | 4 weeks
  Stride length (cm) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.
Step width (centimeter-cm), | 4 weeks
  step width (cm),will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.
Cadence (steps/min) | 4 weeks
  Cadence (steps/min) will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.
step time (second - s) | 4 weeks
  step time ( s) will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.
Stride time (second - s), | 4 weeks
  Stride time (s), will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. The system is comprised of a capacitance-based pressure platform within a treadmill..When the person is standing steadily or on the walking belt, the sensors can receive reactive and normal force measurement in three dimensions with 120Hertz (Hz) frequency. Timing can be monitorized. Temporal and distance recording are taken while the patient is walking and in a static position.

CONTACTS AND LOCATIONS:
Locations (1):
- Fulya Foot Surgery Center, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Feyzioglu O, Ozturk O, Mugrabi S. Effects of custom-made insoles on foot pressure redistribution, gait parameters, and pain in calcaneal apophysitis-a pretest and posttest study. Prosthet Orthot Int. 2021 Dec 1;45(6):532-537. doi: 10.1097/PXR.0000000000000039. PMID 34561380